CLINICAL TRIAL: NCT02709668
Title: Clinical Response and Homocysteine Reduction Using Reduced B-Vitamin Therapy in MTHFR C677T/A1298C Patients With Major Depressive Disorder : an Analysis of Findings
Brief Title: B Vitamins in MTHFR Positive Patients With Major Depression: A Post Hoc Analysis of Findings
Acronym: BVMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: High Point Regional Health Systems (Other)
Responsible Party: Principal Investigator, B. Andrew Farah MD, FAPA, chief of psychiatry high point div. of unc, High Point Regional Health Systems
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AMBFDepression
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: MTHFR depression vitamins Homocysteine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): gel cap with placebo
  Interventions: Other: placebo
- enlyte (Experimental): gel cap of B vitamins brand Enlyte
  Interventions: Dietary Supplement: Enlyte

INTERVENTIONS:
Dietary Supplement: Enlyte — gel cap of reduced B vitamins
  Other Names: reduced B vitamins
  Arms: enlyte
Other: placebo — identical to Enlyte
  Other Names: inert gel cap
  Arms: placebo

SUMMARY:
A randomized double-blind placebo controlled study of reduced B vitamins in patients with major depression who were positive for one or both of the common MTHFR polymorphisms was conducted between 8/1/2014 and 4/3/2015. Homocysteine levels and MADRS scores were used as primary measures. The study was designed to test safety and efficacy of reduced B vitamins in MDD associated with MTHFR. This study examines the data from the trial to see effects, effect sizes, and further, if demographic factors and other patient characteristics correlated with findings.

DETAILED DESCRIPTION:
This original study was designed to evaluate the efficacy and safety of reduced B vitamins as monotherapy in adults with major depressive disorder (MDD) who were also positive for at least 1 methylenetetrahydrofolate reductase (MTHFR) polymorphism associated with depression, and further test the hypothesis that reduced (metabolized) B vitamins will lower homocysteine (HCY) in a majority of clinically responding patients. 330 adult patients with MDD (DSM-5), and positive for MTHFR C677T and/or A1298C polymorphisms were enrolled in a trial conducted between August 1, 2014, and April 3, 2015. 160 patients received placebo, while 170 received a capsule containing a combination of reduced B vitamins. Plasma homocysteine levels were measured at baseline and week 8. The Montgomery-Asberg Depression Rating Scale (MADRS) was used to evaluate efficacy for MDD. This further analysis is conducted on the resultant data, with patient names withheld. It is an extensive look at the findings to determine if response is correlated with HCY reduction and if other factors may be associated with response or non-response.

ELIGIBILITY:
Inclusion Criteria:

* Major depression with MTHFR positive status

Exclusion Criteria:

* dementia, Bipolar, active substance abuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Homocysteine levels | baseline and week 8 of study
  plasma homocysteine levels measured

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | baseline, week 2, week 8
  standard measure of depression

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Mech, MD, Principal Investigator — Mech Healthcare Associates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mech AW, Farah A. Correlation of clinical response with homocysteine reduction during therapy with reduced B vitamins in patients with MDD who are positive for MTHFR C677T or A1298C polymorphism: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2016 May;77(5):668-71. doi: 10.4088/JCP.15m10166. PMID 27035272